CLINICAL TRIAL: NCT00153335
Title: Computerized Risk Assessment in an Employee Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: University of New Mexico (Other)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: CDC-OPHR-R01CD000122; R01CD000122 (NIH)
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2010-02

CONDITIONS: Healthy
Keywords: Health Risk Assessment; Behavior Change; Patient-Provider Interaction; Employee Health; Absenteeism; Tobacco Use; Substance Use; Diet; Exercise; Medication Adherence
MeSH Terms: conditions — Tobacco Use; Substance-Related Disorders; Motor Activity; Medication Adherence

INTERVENTIONS:
Behavioral: patient-provider interaction

SUMMARY:
This is a study to determine whether a computerized risk assessment and focused patient provider interaction can improve health outcomes in an employee population.

DETAILED DESCRIPTION:
The overall goal of the proposed research is to test the effectiveness of a theoretically-based interactive behavioral and health risk assessment system to improve the mental and physical health outcomes of the primary care provided for the adult multicultural members of a university health center-employee-based practice. The new system will include:

1. administration of a computerized behavioral and health risk assessment,
2. calculation of an individualized risk profile for each patient participant,
3. individual patient computerized video training in interaction focused on the risk profile,
4. physician training in patient-provider interaction, motivational interviewing and counseling, and in referral and triage focused on the risk profile, and
5. development of a negotiated care plan between patient and clinician for follow-up care.

Expected outcomes include changes in: risk category scores, utilization patterns, costs for health care services, and health stage of change indicators. Expected impacts (mediating variables) are: compliance with recommendations, health locus of control, differences in patient-provider interaction patterns and patient and clinician satisfaction. If successful, this methodology would contribute significantly to the health promotion goals of Healthy People 2010 and provide much needed evidence of how a behavioral and health risk assessment system can help to reduce ethnic health disparities of multi-cultural populations. This proposal is responsive to CDC's RFA for Health Promotion in the Workplace; in particular it responds to requests for strategy #6: Identification and evaluation of public health informatics and communication strategies and tools to improve health decisions, health alerting, health literacy, or health assessment among employees and employer.

ELIGIBILITY:
Inclusion Criteria:

* Employees who use University of New Mexico providers for medical care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2005-06; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Satisfaction at time of visit
Utilization of health services at one year
Health outcome at one year

SECONDARY OUTCOMES:
Stage of change for health behaviors at one year
Quality of life at one year
Work performance at one year

CONTACTS AND LOCATIONS:
Overall Officials: Deborah L. Helitzer, ScD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Health Sciences Center, Albuquerque, New Mexico, United States